CLINICAL TRIAL: NCT00572897
Title: Study of Fludarabine Based Conditioning for Allogeneic Stem Cell Transplantation for Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0548-00101; P01CA108671-01A2 (NIH); MPD-RC 101 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Myeloproliferative disease; Stem Cell Transplant; Allogeneic Transplant; Conditioning Regimen; Reduced Intensity Regimen; Fludarabine; Melphalan; ATG
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine, Melphalan +/- ATG (Experimental): Fludarabine, Melphalan +/- ATG
  Interventions: Drug: Fludarabine, Melphalan +/- ATG

INTERVENTIONS:
Drug: Fludarabine, Melphalan +/- ATG — Conditioning regimen for Allogenic Stem Cell Transplant:
  Related Donor Fludarabine days -6 to -2 (30mg/m2 IVPB over 30 minutes daily) Melphalan days -3 to -2 (70mg/m2 IVPB over 30 minutes daily)
  Unrelated Donor Fludarabine days -6 to -2 (30mg/m2 IVPB over 30 minutes daily) Melphalan days -3 to -2 (70mg/m2 IVPB over 30 minutes daily) ATG (Thymoglobulin®) days -3 to -1 (0.5 mg/kg IV on day -3 [given over 6 hours], and 2 mg/kg on days -2 and -1 [given over 4 hours])

SUMMARY:
Stem cell transplantation is used to treat may types of diseases. There a 2 types of transplants, conventional (very intense) and reduced intensity-non-myeloablative, also called mini-transplants.

This study proposes to use a conditioning regimen for allogeneic transplantation along with a reduced intensity transplant. Conditioning regiment is the name for the combination of chemotherapy drugs that is given to patients before receiving a transplantation of donor stem cells. It is hoped that the regimen designed for this study proves to be less toxic and has an equal or better anticancer effect than the regimens that are normally used. The regimen being used is a combination of two chemotherapy drugs, fludarabine and melphalan. This regimen has been studied in recipients of matched sibling transplants and in recipients of alternative donor stem cells in other hematologic malignancies. Those subjects, who receive stem cells from an unrelated donor, will also receive and additional drug called ATG or anti thymocyte globulin. ATG suppresses the immune system, thus reducing the chances for the recipient rejecting the transplant (graft).

The purpose of this study is to observe if reduced intensity transplants can be used to allow engraftment or "take" of the donor's bone marrow. Studies conducted in the past show this type of transplant is much less toxic than traditional bone marrow transplants. Reduced intensity transplants may be better tolerated by patients who may experience serious side effects from standard (very intense) stem cell transplant.

The study has been recently amended to follow all subjects for survival.

DETAILED DESCRIPTION:
This study is designed as a single arm Phase II clinical trial in patients with myelofibrosis who are eligible for transplantation from a related donor or from an unrelated donor source. Patients will be accrued into two separate strata defined by donor type. Each of the two strata will be analyzed separately.

Patients will be followed yearly from time of enrollment into the study to assess clinical response and overall, progression and event free survival, as well as incidence and degree of acute and chronic GVHD. We will estimate cumulative survival and transplant related mortality in patients enrolled in each of the two strata.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following disease: Idiopathic myelofibrosis, or spent PV-, or ET-related myelofibrosis in chronic phase (<20% blast cells in the bone marrow) with Lille score >1 at any time, or platelet <100K.
* Age 18-65 years.
* ECOG performance status < 3.
* Life expectancy >3 months.
* Adequate cardiac function, normal LVEF ≥ 45% by MUGA or echocardiogram and adequate pulmonary function DLCO ≥ 50% of predicted.
* Serum creatinine < 1.1 x the upper limit of normal (ULN) or Creatinine Clearance >50 ml/min.
* Serum bilirubin < 2.0 mg/dl, SGPT <2.5 x upper limit of normal
* No evidence of chronic active hepatitis or cirrhosis
* HIV-negative
* Patient is not pregnant
* Patient or guardian able to sign informed consent.
* Patients with >20% myeloblasts in the blood or marrow, extramedullary blast cell proliferation or large foci of blasts in bone marrow biopsy specimens are not eligible.
* Pretransplant splenectomy: MMM patients with variable degrees of splenomegaly, or splenectomized, are eligible to be enrolled. Any decision of having a patient splenectomized prior to transplant will be made in each center prior to enrolling the patient in the study.
* Patients should be off treatment with investigational for at least 4 weeks and have recovered from all toxicities.

Exclusion Criteria:

* Pregnancy
* HIV positive
* > 20% myeloblasts in the peripheral blood or bone marrow
* LVEF < 45%
* DLCO < 50% of predicted
* ECOG performance status ≥ 3
* Chronic active hepatitis or cirrhosis
* Chronic renal insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Giovanni Barosi, MD, Study Chair — Myeloproliferative Disorders-Research Consortium; Damiano Rondelli, MD, Study Chair — Myeloproliferative Disorders-Research Consortium
Locations (12):
- United States (7):
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Ohio State Univesity, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - University of Florence, Florence, IL
  - University of San Martino, San Martino
- Regionala etikprovningsnamnden Goteborg, Gothenburg, Sweden

REFERENCES:
- [Result] Rondelli D, Goldberg JD, Isola L, Price LS, Shore TB, Boyer M, Bacigalupo A, Rambaldi A, Scarano M, Klisovic RB, Gupta V, Andreasson B, Mascarenhas J, Wetzler M, Vannucchi AM, Prchal JT, Najfeld V, Orazi A, Weinberg RS, Miller C, Barosi G, Silverman LR, Prosperini G, Marchioli R, Hoffman R. MPD-RC 101 prospective study of reduced-intensity allogeneic hematopoietic stem cell transplantation in patients with myelofibrosis. Blood. 2014 Aug 14;124(7):1183-91. doi: 10.1182/blood-2014-04-572545. Epub 2014 Jun 24. PMID 24963042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 2007 to 2011 at 11 centers affiliated with the Myeloproliferative Disorders Research Consortium (MPD-RC)
Groups:
- Sibling Donor: Patients received a stem cell transplant from sibling
- Unrelated Donor: Patients received a stem cell transplant from an unrelated donor
Period: Overall Study
Arm/Group | Sibling Donor | Unrelated Donor
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with myelofibrosis who received a stem cell transplant from either a sibling or unrelated donor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sibling Donor | Unrelated Donor | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Median (Full Range); unit: years] — Median age at the time of transplant
  years | 55 [40 to 65] | 56 [30 to 65] | 55 [30 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 19 | 19 | 38
Diagnosis [Number; unit: participants] — Primary Myelofibrosis (PMF); Post-Polycythemia vera (PV-MF); Post-Essential Thrombocythemia (ET-MF)
  participants
    PMF | 14 | 25 | 39
    PV-MF | 3 | 5 | 8
    ET-MF | 15 | 4 | 19
Lille score [Number; unit: participants] — The Lille scoring system was created by Dupriez and coworkers and used in selecting intermediate- and higher-risk patients as candidates for Autologous Stem Cell Transplant (ASCT). A platelet count of >100 × 109/L in patients with IM was associated with an adverse outcome and created a complete blood count scoring system using three parameters: Hgb < 10 gm/dL; WBC < 4 or > 30 × 109/L; and platelet count <100 × 109/L. Each event was given a score of 1. Higher scores indicate lower median survival.
  participants
    0 | 3 | 0 | 3
    1 | 20 | 23 | 43
    2 | 9 | 11 | 20
Patient: donor gender [Number; unit: participants]
  Female:Female | 6 | 7 | 13
  Male:Male | 7 | 8 | 15
  Male:Female | 10 | 6 | 16
  Female:Male | 9 | 13 | 22
JAK-2V617F [Number; unit: participants]
  Positive | 12 | 18 | 30
  Negative | 17 | 16 | 33
  Unknown | 3 | 0 | 3
Bone Marrow Fibrosis [Number; unit: participants] — European consensus on grading bone marrow fibrosis:
  MF - 0 Scattered linear reticulin with no intersections (cross-overs) corresponding to normal bone marrow; MF - 1 Loose network of reticulin with many intersections, especially in perivascular areas; MF - 2 Diffuse and dense increase in reticulin with extensive intersections,occasionally with only focal bundles of collagen and/or focal osteosclerosis; MF - 3 Diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis
  participants
    Grade 1 | 0 | 2 | 2
    Grade 2 | 2 | 6 | 8
    Grade 3 | 18 | 23 | 41
    Unknown | 12 | 3 | 15
Splenomegaly [Number; unit: participants]
  Yes | 24 | 28 | 52
  No | 3 | 1 | 4
  Splenectomy | 5 | 5 | 10
Karyotype [Number; unit: participants]
  Normal | 14 | 14 | 28
  One abnormality | 7 | 9 | 16
  Complex abnormality | 5 | 0 | 5
  Unknown | 6 | 11 | 17
Stem cell source [Number; unit: participants]
  Peripheral blood | 26 | 31 | 57
  Bone Marrow | 6 | 3 | 9
HLA match [Number; unit: participants]
  Full HLA matched | 30 | 25 | 55
  HLA 1 Ag mismatched, no allele mismatched | 2 | 4 | 6
  HLA Ag matched, 1 0r 2 alleles mismatched | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is Progression-free Survival.
Description: Number of participants alive at 2 years who are progression-free
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 32 | 34
participants | 24 | 11

2. Secondary Outcome: Response Outcomes
Description: assessed according to the IWG Criteria
Time Frame: 180 days
Population: Clinical responses were assessed according to the IWG-MRT 2006 criteria in 46 patients (29 sibling and 17 unrelated transplants) who survived at least 180 days.
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 29 | 17
participants
  clinical complete response | 7 | 6
  clinical partial response | 8 | 1
  clinical improvement | 11 | 5
  stable disease | 2 | 4
  progressive disease | 0 | 1

3. Secondary Outcome: Overall Survival
Description: The number of patients alive at last follow-up.
Time Frame: 73 months
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 32 | 34
participants | 25 | 11

4. Secondary Outcome: Absolute Neutrophil Count (ANC)
Description: Patients with ANC ≥0.5 × 10^9/L
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 32 | 34
participants
  yes | 31 | 26
  no | 1 | 8

5. Secondary Outcome: PLT
Description: Patients with PLT ≥20 × 109/L
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 32 | 34
participants
  yes | 28 | 20
  no | 4 | 14

6. Secondary Outcome: Transplant-related Mortality
Description: Transplant-related Mortality including Graft-versus-host disease (GVHD)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 32 | 34
participants
  yes | 3 | 20
  no | 29 | 14

ADVERSE EVENTS:
Description: all adverse events reported under serious adverse events. other non-serious adverse events were not separated out.
Arm/Group | Sibling Donor | Unrelated Donor
Serious Adverse Events (participants affected / at risk) | 8/32 | 23/34
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sibling Donor (N=32) | Unrelated Donor (N=34)
Death (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — Progression of disease
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Secondary malignancy
Death (Immune system disorders) | 3 (3) | 5 (5) — acute graft-versus-host disease (aGVHD)
Death (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — hemorrhage
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Respiratory failure
Death (Cardiac disorders) | 1 (1) | 0 (0) — Heart Failure
Death (Surgical and medical procedures) | 0 (0) | 20 (20) — Transplant-related complications
Death (Renal and urinary disorders) | 0 (0) | 2 (2) — Renal Failure
Death (Vascular disorders) | 0 (0) | 1 (1) — Venous occlusive disease
Death (Infections and infestations) | 0 (0) | 1 (1) — Viral infection
Death (Surgical and medical procedures) | 0 (0) | 1 (1) — Event secondary to graft failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No